CLINICAL TRIAL: NCT06838468
Title: Detection of Advanced Chronic Liver Disease in Patients With Alcohol Use Disorder in the Hospital Detoxification Unit
Brief Title: cACLD in Patients With Alcohol Use Disorder in the Hospital Detoxification Unit
Acronym: HEP-UHD
Status: Enrolling by invitation | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jordi Sanchez-Delgado, Head of the hepatology hospitalization unit, Corporacion Parc Tauli
Other Study IDs: 2024/5057; 2024/5057 (Other: CEIM Parc Tauli)
Record Dates: First submitted 2025-01-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Liver Disease Chronic; Cirrhosis; Detoxification; Alcohol Abuse/Dependence
Keywords: chronic advance liver disease; detoxification unit; elastography; liver risk score
MeSH Terms: conditions — Fibrosis; Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with excessive alcohol consumption admitted to the hospital detoxification unit: The intervention performed on patients who have been electively admitted to the hospital detoxification unit consists of diagnostic tests to assess potential liver damage secondary to alcohol consumption. These are usually young patients with very high alcohol intake who, under normal circumstances, would need to be evaluated on an outpatient basis. Since the potential prevalence of advanced liver disease is expected to be higher in this subgroup of patients, the hospital stay is utilized to carry out all these tests quickly. The tests performed will include a general blood analysis to evaluate liver and kidney function, an assessment of the prevalence of metabolic diseases such as obesity, hypertension, or diabetes, an abdominal ultrasound, and elastography to assess liver stiffness.
  Interventions: Diagnostic Test: Screening of compensated advance chronic liver disease

INTERVENTIONS:
Diagnostic Test: Screening of compensated advance chronic liver disease — The tests performed will include a general blood analysis to evaluate liver and kidney function, an assessment of the prevalence of metabolic diseases such as obesity, hypertension, or diabetes, an abdominal ultrasound, and elastography to assess liver stiffness.
  Another intervention to be studied is whether the request for diagnostic tests to evaluate liver disease, as well as the visit of the hepatologist during hospitalization in the detoxification unit, influences subsequent alcohol abstinence. To this end, abstinence will be assessed six months after admission to the alcohol detoxification unit and compared with a retrospective cohort of patients admitted to the detoxification unit one year ago, in whom no liver disease evaluation was conducted neither information of potencial liver damage was offered by hepatologist and the intervention was carried out only by the psychiatrists responsible for the unit.

SUMMARY:
The aim of this study is to conduct a quick assessment of potential liver damage caused by chronic alcohol consumption. Taking advantage of the patient's admission to a specialized detoxification unit, several tests will be performed to determine the extent of liver damage through blood tests, ultrasound, and FibroScan

DETAILED DESCRIPTION:
There is very little recent data on the prevalence of advance chronic liver disease in high-risk patients, particularly in our region, making studies evaluating this necessary.

In the European clinical practice guidelines (EASL Clinical Practice Guidelines: Management of Alcohol-Related Liver Disease), it is recommended to screen for advance chronic liver disease in high-risk populations such as patients in rehabilitation and detox clinics and heavy drinkers. advance chronic liver disease should be considered in patients presenting with extrahepatic manifestations of alcohol use disorder, such as peripheral symmetric neuropathy, pancreatitis, and cardiomyopathy, among others.

Screening for liver disease in high-risk groups should not only include liver function tests (e.g., gamma-glutamyl transferase [GGT], alanine aminotransferase [ALT], or aspartate aminotransferase [AST]) but also include testing for liver fibrosis (e.g., transient elastography such as FibroScan®), given that advanced liver disease may occur in patients with normal liver profiles.

If any abnormalities are detected in liver profiles or elastography, an abdominal ultrasound should be performed to rule out hepatocellular carcinoma and a complete liver disease study should be carried out to exclude alternative or additional causes of liver damage. Current clinical guidelines (Spanish, European, and American) do not specify which tools to use in each risk subgroup.

The primary objective is to assess the prevalence of advance chronic liver disease measured by transient elastography in patients admitted to the Hospital Detoxification Unit and the acute psychiatric unit with dual pathology and harmful alcohol consumption.

This is a prospective, descriptive, single-center study conducted at Hospital Parc Taulí in Sabadell on patients admitted to the Hospital Detoxification Unit and the psychiatric unit with a diagnosis of dual pathology and harmful alcohol consumption. The study duration will be one year (from June 2024 to June 2025).

We will obtein clinical Variables like date of birth, sex, ethnicity, height, height, medical history (e.g., diagnosis of diabetes, dyslipidemia, hypertension, or underlying psychiatric disorder); Laboratory Variables: ALT, AST, alkaline phosphatase (ALP), GGT, total bilirubin, INR, platelets, glucose, HbA1c, total cholesterol, HDL, LDL, TSH, ferritin, and transferrin saturation. For patients with abnormal liver profiles, a second etiological study will be performed, including ceruloplasmin, copper, alpha-1 antitrypsin, ANA and SLA autoantibodies, immunoglobulins (IgA, IgG, IgM), and protein electrophoresis.

Elastography Variables: FibroScan® values and CAP (Control Attenuation Parameter) to estimate liver stiffness and quantify hepatic fat, respectively.

Radiological Variables: Abdominal ultrasound findings (e.g., homogeneous or heterogeneous liver, presence of steatosis, nodular liver borders, splenomegaly, recanalization of the paraumbilical vein, collateral circulation, portal velocity, hepatic nodules). Endoscopic Variables: For patients diagnosed with advance chronic liver disease, esophagogastroduodenoscopy will be performed to rule out esophageal varices if criteria are met. Serological Variables for Fibrosis Estimation: LiverRisk score, APRI, FIB-4, Forns index, AAR (AST to ALT ratio).

Regardless of liver profile abnormalities, an abdominal ultrasound will be requested to evaluate parenchymal changes and other indirect signs of liver disease and/or portal hypertension. Additional data collected by psychiatry will include the patient's date of birth, years of alcohol consumption, grams of alcohol/day measured in Standard Drink Units (SDUs), weight, height, relevant cardiovascular diseases (hypertension, diabetes, dyslipidemia), and underlying psychiatric disorders.

A hepatology consultation will be requested, and FibroScan® will be performed during hospitalization. All fibrosis scores (LiverRisk score, APRI, FIB-4, Forns, and AAR) will be calculated using demographic and laboratory data.

If liver profile abnormalities are detected upon admission, a complete second etiological study will be requested.

All patients, regardless of whether they have advanced chronic liver disease or not, will be evaluated by a hepatologist who will provide information about the results of the diagnostic tests performed and the potential harmful effects of alcohol on the liver and overall health. This will reinforce the information provided by the psychiatrist in an effort to encourage the patient to cease alcohol consumption.

If the patient presents advance chronic liver disease (FibroScan® >8 KPa) or analytical, elastographic, or radiological evidence suggestive of cirrhosis will be referred to hepatology outpatient clinics for further evaluation and follow-up. Patients without advance chronic liver disease findings will be referred to primary care by their attending psychiatrist for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the detoxification unit for alcohol use disorder
* Patients admitted to the psychiatry unit for dual pathology with harmful alcohol consumption (> 30 g/day in men (3 standard drinks) and > 20 g/day in women (2 standard drinks))

Exclusion Criteria:

* Refusal to undergo additional tests (blood analysis, ultrasound, and FibroScan)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the detoxification unit for alcohol use disorder or de psychiatry unit for dual pathology with harmful alcohol consumption
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of advanced chronic liver disease in patients who are electively admitted to the hospital alcohol detoxification unit | 5 days
  Prevalence of pathological findings in the fibroscan that suggest compensated chronic liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sánchez Delgado, MD. PhD, Principal Investigator — Consorci Corporació Sanitària Parc Taulí
Locations (1):
- Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Information about the project will be shared if another center is interested in participating and conducting a multicenter study
Supporting Information: SAP
Time Frame: The information will be available at the end of the study in January 2026
Access Criteria: Other researchers will have the opportunity to contact the principal investigator of the study and discuss any rellevant study information

REFERENCES:
- [Result] Serra-Burriel M, Juanola A, Serra-Burriel F, Thiele M, Graupera I, Pose E, Pera G, Grgurevic I, Caballeria L, Piano S, van Kleef L, Reichert M, Roulot D, Pericas JM, Schattenberg JM, Tsochatztis EA, Guha IN, Garcia-Retortillo M, Hernandez R, Hoyo J, Fuentes M, Exposito C, Martinez A, Such P, Madir A, Detlefsen S, Tonon M, Martini A, Ma AT, Pich J, Bonfill E, Juan M, Soria A, Carol M, Gratacos-Gines J, Morillas RM, Toran P, Navarrete JM, Torrejon A, Fournier C, Llorca A, Arslanow A, de Koning HJ, Cucchietti F, Manns M, Newsome PN, Hernaez R, Allen A, Angeli P, de Knegt RJ, Karlsen TH, Galle P, Wong VW, Fabrellas N, Castera L, Krag A, Lammert F, Kamath PS, Gines P; LiverScreen Consortium Investigators. Development, validation, and prognostic evaluation of a risk score for long-term liver-related outcomes in the general population: a multicohort study. Lancet. 2023 Sep 16;402(10406):988-996. doi: 10.1016/S0140-6736(23)01174-1. Epub 2023 Aug 9. PMID 37572680
- [Result] Crabb DW, Bataller R, Chalasani NP, Kamath PS, Lucey M, Mathurin P, McClain C, McCullough A, Mitchell MC, Morgan TR, Nagy L, Radaeva S, Sanyal A, Shah V, Szabo G; NIAAA Alcoholic Hepatitis Consortia. Standard Definitions and Common Data Elements for Clinical Trials in Patients With Alcoholic Hepatitis: Recommendation From the NIAAA Alcoholic Hepatitis Consortia. Gastroenterology. 2016 Apr;150(4):785-90. doi: 10.1053/j.gastro.2016.02.042. Epub 2016 Feb 24. No abstract available. PMID 26921783
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of alcohol-related liver disease. J Hepatol. 2018 Jul;69(1):154-181. doi: 10.1016/j.jhep.2018.03.018. Epub 2018 Apr 5. No abstract available. PMID 29628280
- [Result] Addolorato G, Mirijello A, Leggio L, Ferrulli A, D'Angelo C, Vassallo G, Cossari A, Gasbarrini G, Landolfi R, Agnes S, Gasbarrini A; Gemelli OLT Group. Liver transplantation in alcoholic patients: impact of an alcohol addiction unit within a liver transplant center. Alcohol Clin Exp Res. 2013 Sep;37(9):1601-8. doi: 10.1111/acer.12117. Epub 2013 Apr 11. PMID 23578009
- [Result] Askgaard G, Leon DA, Kjaer MS, Deleuran T, Gerds TA, Tolstrup JS. Risk for alcoholic liver cirrhosis after an initial hospital contact with alcohol problems: A nationwide prospective cohort study. Hepatology. 2017 Mar;65(3):929-937. doi: 10.1002/hep.28943. Epub 2017 Jan 6. PMID 27862159
- [Result] Rehm J, Taylor B, Mohapatra S, Irving H, Baliunas D, Patra J, Roerecke M. Alcohol as a risk factor for liver cirrhosis: a systematic review and meta-analysis. Drug Alcohol Rev. 2010 Jul;29(4):437-45. doi: 10.1111/j.1465-3362.2009.00153.x. PMID 20636661
- [Result] Gines P, Krag A, Abraldes JG, Sola E, Fabrellas N, Kamath PS. Liver cirrhosis. Lancet. 2021 Oct 9;398(10308):1359-1376. doi: 10.1016/S0140-6736(21)01374-X. Epub 2021 Sep 17. PMID 34543610
- [Result] Passi S, Rothschild-Boros MC, Fasella P, Nazzaro-Porro M, Whitehouse D. An application of high performance liquid chromatography to analysis of lipids in archaeological samples. J Lipid Res. 1981 Jul;22(5):778-84. PMID 7026710